CLINICAL TRIAL: NCT03178851
Title: A Phase Ib Study Evaluating Cobimetinib Plus Atezolizumab in Patients With Advanced BRAF V600 Wild-Type Melanoma Who Have Progressed During or After Treatment With Anti-PD-1 Therapy and Atezolizumab Monotherapy in Patients With Previously Untreated Advanced BRAF V600 Wild-Type Melanoma
Brief Title: Cobimetinib (Targeted Therapy) Plus Atezolizumab (Immunotherapy) in Participants With Advanced Melanoma Whose Cancer Has Worsened During or After Treatment With Previous Immunotherapy and Atezolizumab Monotherapy in Participants With Previously Untreated Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO39721; 2016-004402-34 (EudraCT Number)
Record Dates: First submitted 2017-06-01; First posted 2017-06-07 (Actual); Results first posted 2020-06-12 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — atezolizumab; cobimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A (Experimental): Participants with disease progression on or after treatment with an anti-PD-1 agent will receive cobimetinib and atezolizumab treatment during 28-day cycles.
  Interventions: Biological: Atezolizumab; Drug: Cobimetinib
- Cohort B (Experimental): Participants with disease progression on or after treatment with an anti-PD-1 agent will receive cobimetinib prior to initiating atezolizumab treatment during Cycle 1. During subsequent 28-day cycles participants will initiate both atezolizumab and cobimetinib on Day 1 of each cycle. Participants in this cohort will undergo tumor biopsies before and during treatment.
  Interventions: Drug: Cobimetinib; Biological: Atezolizumab
- Cohort C (Experimental): Participants with advanced melanoma, who have not received previous treatment, will receive atezolizumab monotherapy during 21-day cycles.
  Interventions: Biological: Atezolizumab

INTERVENTIONS:
Biological: Atezolizumab — Atezolizumab, 840 mg intravenously every two weeks (Q2W) on Days 1 and 15 of each 28-day cycle, until loss of clinical benefit
  Other Names: Tecentriq
  Arms: Cohort A
Drug: Cobimetinib — Cobimetinib, 60 mg orally once daily (QD) on Days 1-21 of each 28-day cycle, until loss of clinical benefit
  Other Names: Cotellic
  Arms: Cohort A; Cohort B
Biological: Atezolizumab — Atezolizumab, 840 mg intravenously on Day 15 of Cycle 1; thereafter Q2W on Days 1 and 15 of Cycle 2 and all subsequent 28-day cycles, until loss of clinical benefit
  Other Names: Tecentriq
  Arms: Cohort B
Biological: Atezolizumab — Atezolizumab, 1200 mg intravenously every three weeks (Q3W) on Day 1 of each 21-day cycle, until loss of clinical benefit
  Other Names: Tecentriq
  Arms: Cohort C

SUMMARY:
This study will evaluate the preliminary efficacy, safety, and pharmacokinetics of cobimetinib and atezolizumab in participants with advanced BRAF V600-wild type (WT), metastatic, or unresectable locally advanced melanoma who have progressed on prior anti-PD-1 therapy. In addition, this study will evaluate the efficacy, safety, and pharmacokinetics of atezolizumab monotherapy in participants with BRAFV600-WT metastatic or unresectable locally advanced melanoma, who have not been previously treated.

ELIGIBILITY:
Inclusion criteria

Disease-Specific Inclusion Criteria: Cohorts A and B:

* Histologically confirmed Stage IV (metastatic) or unresectable Stage IIIc BRAF V600 WT (locally advanced) melanoma
* Documentation of BRAF V600 mutation-negative status in melanoma tumor tissue (archival [< 5 years old] or newly obtained) through use of a clinical mutation test approved by the local health authority
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Disease progression on or after treatment with a programmed death (PD)-1 inhibitor either as monotherapy or in combination with other agent(s)

Additional Disease-Specific Inclusion Criteria in Cohort B (Biopsy Cohort):

* Progressed on or after anti-PD-1 therapy within 12 weeks before study start
* Received a minimum of two cycles of anti-PD-1 therapy
* Meet the following criteria for resistance to an anti-PD-1 agent: primary resistance defined as disease progression, according to RECIST v1.1, as best response; secondary resistance defined as disease progression after initial confirmed response according to RECIST v1.1
* Consent to undergo tumor biopsies of accessible lesions, before and during treatment and at radiographic progression, for biomarker analyses.
* Have at least two accessible lesions that are amenable to excisional or core-needle (minimum three cores and minimum diameter 18 gauge; however, 16 gauge is desirable) biopsy without unacceptable risk of a major procedural complication. Exceptions may be made if patient has only one lesion that allows multiple biopsies.

Disease-Specific Inclusion Criteria: Cohort C:

* Histologically confirmed Stage IV (metastatic) or unresectable Stage IIIc BRAFV600-WT (locally advanced) melanoma
* Naive to prior systemic anti-cancer therapy for melanoma
* Documentation of BRAFV600 mutation-negative status in melanoma tumor tissue (archival [< 5 years old] or newly obtained) through use of a clinical mutation test approved by the local health authority
* A representative, formalin-fixed, paraffin-embedded (FFPE) tumor specimen in a paraffin block (preferred) or 20 slides containing unstained, freshly cut, serial sections must be submitted along with an associated pathology report prior to study entry.
* Measurable disease according to RECIST v1.1.

General Inclusion Criteria:

* Ability to comply with the study protocol, in the investigator's judgment
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Available and adequate baseline tumor tissue sample
* Life expectancy ≥ 18 weeks
* Adequate hematologic and end-organ function, defined by laboratory test results, obtained within 14 days before initiation of study treatment
* For women of childbearing potential: abstinent or use an effective form of contraceptive method for at least 3 months for cobimetinib and at least 5 months for atezolizumab. Women must refrain from donating eggs during this same period.
* For men: abstinent or use contraceptive measures and agreement to refrain from donating sperm for at least 3 months after cobimetinib and atezolizumab

Exclusion criteria

* Prior treatment with a mitogen activated-protein kinase (MAPK) inhibitor
* Ocular melanoma
* Major surgical procedure other than for diagnosis within 4 weeks before initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study
* Traumatic injury within 2 weeks before initiation of study treatment
* Palliative radiotherapy within 14 days before initiation of study treatment
* Active malignancy (other than BRAF V600 mutation-negative melanoma) or malignancy within 3 years
* Treatment with any anti-cancer agent 14 days prior to Cycle, Day 1 other than aPD-1 based therapy
* Adverse events from prior anti-cancer therapy that have not resolved to Grade ≤ 1. Clinically stable patients with manageable immune-related adverse events resulting from prior cancer immunotherapy may be eligible for the study.
* For Cohort C only: any prior anti-cancer therapy for advanced melanoma
* History or evidence of ongoing serous retinopathy or retinal vein occlusion (RVO) at baseline
* History of clinically significant cardiac dysfunction
* Active or untreated central nervous system (CNS) metastases
* History of metastases to brain stem, midbrain, pons, or medulla, or within 10 millimeter (mm) of the optic apparatus (optic nerves and chiasm)
* History of leptomeningeal metastatic disease
* Human immunodeficiency virus (HIV) infection
* Active tuberculosis
* Severe infection within 4 weeks before initiation of study treatment
* Signs or symptoms of infection within 2 weeks before initiation of study treatment
* Treatment with oral or intravenous (IV) antibiotics within 2 weeks prior to Day 1 of Cycle 1
* Active or chronic viral hepatitis B or C infection
* Active or history of autoimmune disease or immune deficiency
* Prior allogeneic stem cell or solid organ transplantation
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Treatment with systemic immunosuppressive medications with the following exceptions:
* Patients who have received acute, low-dose systemic immunosuppressant medication (≤ 10 mg/day oral prednisone or equivalent) or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Medical Monitor approval has been obtained.
* Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Current severe, uncontrolled systemic disease other than cancer
* Any Grade >/=3 hemorrhage or bleeding event within 28 days of Day 1 of Cycle 1
* History of stroke, reversible ischemic neurological defect, or transient ischemic attack within 6 months prior to Day 1
* Anticipated use of any concomitant medication during or within 7 days before initiation of study treatment that is known to cause QT prolongation
* Any psychological, familial, sociological, or geographic condition that may hamper compliance with the protocol and follow-up after treatment discontinuation
* History of malabsorption or other clinically significant metabolic dysfunction that may interfere with absorption of oral study treatment
* Pregnant or breastfeeding, or intending to become pregnant during the study
* Known clinically significant liver disease
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the participant at high risk for treatment complications
* Treatment with a live, attenuated vaccine within 4 weeks before initiation of study treatment, or anticipation of need for such a vaccine during the course of the study
* Known hypersensitivity to any component of the atezolizumab or cobimetinib formulations
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Treatment with any other investigational agent or participation in another clinical study with therapeutic intent
* Inability or unwillingness to swallow pills
* Requirement for concomitant therapy or food that is prohibited during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2020-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (43):
- United States (6):
  - HonorHealth Research Institute - Bisgrove, Scottsdale, Arizona
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
- Australia (7):
  - Blacktown Hospital, Blacktown, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Mid North Coast Cancer Institute, Port Macquarie, New South Wales
  - Greenslopes Private Hospital; Clinic Pharmacy, Greenslopes, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - University Clinic Ctr Sarajevo, Sarajevo
- Brazil (7):
  - Instituto de Ensino e Pesquisa Clinica do Ceara, Fortaleza, Ceará
  - Cenantron - Centro Avancado de Tratamento Oncologico, Belo Horizonte, Minas Gerais
  - Instituto Nacional de Cancer - INCa; Oncologia, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
- South Africa (7):
  - Cape Town Oncology Trials, Cape Town
  - GVI Constantiaberg, Cape Town
  - Johese Clinical Research, Centurion
  - Cancercare, George
  - Wits Clinical Research; Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg
  - Cancercare, Port Elizabeth
  - Steve Biko Academic Hospital; Oncology, Pretoria
- Spain (9):
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela, LA Coruña
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramón y Cajal; Pharmacy, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Hospital Universitario La Paz; Servicio de Oncologia, Madrid
- Ukraine (5):
  - Central Municipal Hospital - Uzhgorod State University, Uzhhorod, Chernihiv Governorate
  - Public Institution: City Multispecialty Clinical Hospital #4 under Dnipropetrovsk Regional Council, Dnipropetrovsk
  - National Cancer Institute MOH of Ukraine, Kiev
  - Lviv State Oncology Regional Treatment and Diagnostic Centre, Lviv
  - Sumy Regional Clinical Onc Ctr, Sumy

REFERENCES:
- [Derived] Sandhu S, Atkinson V, Cao MG, Medina T, Rivas AS, Menzies AM, Caro I, Roberts L, Song Y, Yan Y, Guo Y, Xue C, Long GV. Phase 1b study of cobimetinib plus atezolizumab in patients with advanced BRAFV600 wild-type melanoma progressing on prior anti-programmed death-1 therapy. Eur J Cancer. 2023 Jan;178:180-190. doi: 10.1016/j.ejca.2022.10.019. Epub 2022 Nov 2. PMID 36455412
- [Derived] Barteselli G, Goodman GR, Patel Y, Caro I, Xue C, McCallum S. Characterization of Serous Retinopathy Associated with Cobimetinib: Integrated Safety Analysis of Four Studies. Drug Saf. 2022 Dec;45(12):1491-1499. doi: 10.1007/s40264-022-01248-2. Epub 2022 Oct 30. PMID 36310331
- [Derived] de Azevedo SJ, de Melo AC, Roberts L, Caro I, Xue C, Wainstein A. First-line atezolizumab monotherapy in patients with advanced BRAFV600 wild-type melanoma. Pigment Cell Melanoma Res. 2021 Sep;34(5):973-977. doi: 10.1111/pcmr.12960. Epub 2021 Feb 15. PMID 33476492

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Participants with disease progression on or after treatment with an anti-PD-1 agent initiated dosing with atezolizumab concurrently with cobimetinib. Participants received intravenous (IV) atezolizumab every two weeks (Q2W) on Days 1 and 15 of all cycles. Participants received oral cobimetinib once daily (QD) on Days 1-21 of each 28-day cycle.
- Cohort B: Participants with disease progression on or after treatment with an anti-PD-1 agent received cobimetinib prior to initiating IV atezolizumab treatment on Day 15 of Cycle 1. Participants continued to receive atezolizumab on Days 1 and 15 from Cycle 2 onwards. Oral cobimetinib was given QD on Days 1-21 of each 28-day cycle. Participants in this cohort underwent tumor biopsies before and during treatment.
- Cohort C: Participants with advanced melanoma, who had not received previous treatment, received IV atezolizumab monotherapy every 3 weeks (Q3W).
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 92 | 11 | 52
Completed | 0 | 0 | 0
Not Completed | 92 | 11 | 52
Not completed — Death | 48 | 2 | 25
Not completed — Withdrawal by Subject | 8 | 0 | 0
Not completed — Lost to Follow-up | 5 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Study Termination by Sponsor | 31 | 7 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 92 | 11 | 52 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (11.8) | 62.3 (9.6) | 61.2 (11.8) | 61.0 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 3 | 17 | 53
  Male | 59 | 8 | 35 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 25 | 32
  Not Hispanic or Latino | 82 | 10 | 26 | 118
  Unknown or Not Reported | 4 | 0 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 4 | 5
  White | 88 | 11 | 46 | 145
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Investigator-Assessed Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with confirmed objective response (OR). Confirmed OR is defined as complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 92 | 11 | 52
Percentage of Participants | 12.0 [6.12 to 20.39] | 36.4 [10.93 to 69.21] | 38.5 [25.30 to 52.98]

2. Primary Outcome: Investigator-Assessed Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with CR, PR, or stable disease (SD) at 16 weeks. Per RECIST v1.1, CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum on study. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline, or the appearance of one or more new lesions.
Time Frame: Week 16
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 92 | 11 | 52
Percentage of Participants | 37.0 [27.12 to 47.66] | 54.5 [23.38 to 83.25] | 46.2 [32.23 to 60.53]

3. Secondary Outcome: Investigator-Assessed Duration of Response (DOR)
Description: DOR is defined as the time from the first occurrence of documented OR to disease progression, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: Up to approximately 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 92 | 11 | 52
Months | 24.2 [7.4 to 24.2] | NA [7.8 to NA] — Value is not available due to an insufficient number of participants with the event. | NA [20.1 to NA] — Value is not available due to an insufficient number of participants with the event.

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from Cycle 1, Day 1 to death from any cause.
Time Frame: Up to approximately 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 92 | 11 | 52
Months | 12.5 [9.4 to 16.7] | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event. | 22.0 [11.7 to NA] — Value is not available due to an insufficient number of participants with the event.

5. Secondary Outcome: Investigator-Assessed Progression-Free Survival (PFS)
Description: PFS is defined as the time from Cycle 1, Day 1 to the first occurrence of disease progression, as determined by the investigator according to RECIST v1.1, or death from any cause, whichever occurs first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: Up to approximately 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 92 | 11 | 52
Months | 3.7 [3.5 to 5.6] | 9.3 [1.8 to 20.1] | 3.7 [2.1 to 7.4]

6. Secondary Outcome: Serum Concentration of Atezolizumab
Time Frame: Cycle 1, Day 15; Day 1 of Cycles 2, 3, 4, 8
Population: Pharmacokinetic (PK) analyses were performed on all participants that received at least one dose of study drug and who had at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 92 | 11 | 52
ug/mL
  Cmax - Cycle 1 Day 15: number analyzed (Participants) | 91 | 11 | 52
  Cmax - Cycle 1 Day 15 | 271 (22.1) | 275 (21.9) | 388 (20.5)
  Cmin - Cycle 2 Day 1: number analyzed (Participants) | 91 | 11 | 52
  Cmin - Cycle 2 Day 1 | 65.3 (330) | 32.9 (1540) | 73.2 (55.0)
  Cmin - Cycle 3 Day 1: number analyzed (Participants) | 91 | 11 | 52
  Cmin - Cycle 3 Day 1 | 92.4 (442) | 37.6 (7490) | 113 (47.8)
  Cmin - Cycle 4 Day 1: number analyzed (Participants) | 91 | 11 | 52
  Cmin - Cycle 4 Day 1 | 121 (237) | 83.7 (844) | 128 (50.8)
  Cmin - Cycle 8 Day 1: number analyzed (Participants) | 91 | 11 | 52
  Cmin - Cycle 8 Day 1 | 210 (46.8) | NA (NA) — Value unavailable due to insufficient number of evaulable samples. | 159 (58.7)

7. Secondary Outcome: Plasma Concentration of Cobimetinib
Time Frame: Cycle 1, Day 15
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 92 | 11
ug/mL
  Cycle 1 Day 15 - Ctrough: number analyzed (Participants) | 90 | 8
  Cycle 1 Day 15 - Ctrough | 165 (137) | 125 (86.6)
  Cycle 1 Day 15 - Css: number analyzed (Participants) | 90 | 8
  Cycle 1 Day 15 - Css | 318 (75.2) | 208 (59.6)

8. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline through follow up
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 92 | 11 | 52
Percentage of Participants | 98.9 | 100 | 100

9. Secondary Outcome: Change From Baseline in Percentage of Participants With Anti-drug Antibodies (ADAs) to Atezolizumab
Description: To evaluate the immune response to atezolizumab the percentage of participants with ADAs to atezolizumab will be determined at baseline and during the study.
Time Frame: Cycle 1 Day 1 pre-dose to 120 days after the last dose of study medication
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 92 | 11 | 52
Percentage of Participants | 32.5 | 30.0 | 10.0

10. Secondary Outcome: Cohort C: Independent-Review-Committee-Assessed (IRC) ORR
Description: ORR is defined as the percentage of participants with confirmed objective response (OR), as determined by an independent review committee (IRC) according to RECIST v1.1. Confirmed OR is defined as complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart, as determined by an independent review committee (IRC) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: Approximately 2 years for Cohorts A and B and 19 months for Cohort C
Population: The analysis populations included all participants with measureable disease at baseline as measured by either the investigator or by an IRC.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort C
Number analyzed (Participants) | 44
Percentage of Participants | 27.3 [14.96 to 42.79]

11. Secondary Outcome: Cohort C: IRC-Assessed DCR
Description: DCR is defined as the percentage of participants with CR, PR, or stable disease (SD), as determined by an independent review committee (IRC) according to RECIST v1.1. CR is defined as disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression, taking as reference the smallest sum on study. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline, or the appearance of one or more new lesions.
Time Frame: Approximately 21 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort C
Number analyzed (Participants) | 44
Percentage of Participants | 38.6 [24.36 to 54.50]

12. Secondary Outcome: Cohort C: IRC-Assessed DOR
Description: DOR is defined as the time from the first occurrence of documented OR to disease progression, as determined by an independent review committee (IRC) according to RECIST v1.1, or death from any cause, whichever occurs first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: Approximately 21 months
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort C
Number analyzed (Participants) | 52
Months | NA [NA to NA] — Value is not available due to an insufficient number of participants with the event.

13. Secondary Outcome: Cohort C: IRC-Assessed PFS
Description: PFS is defined as the time from Cycle 1, Day 1 to the first occurrence of disease progression, as determined by an independent review committee (IRC) according to RECIST v1.1, or death from any cause, whichever occurs first. Disease progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study including baseline; or the appearance of one or more new lesions.
Time Frame: Approximately 21 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort C
Number analyzed (Participants) | 52
Months | 3.7 [2.1 to 11.7]

ADVERSE EVENTS:
Time Frame: Baseline through follow up
Arm/Group | Cohort A | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 48/92 | 2/11 | 25/52
Serious Adverse Events (participants affected / at risk) | 42/92 | 5/11 | 15/52
Other Adverse Events (participants affected / at risk) | 90/92 | 11/11 | 50/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=92) | Cohort B (N=11) | Cohort C (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartase aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 1 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Angiogram (Investigations) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=92) | Cohort B (N=11) | Cohort C (N=52)
Anaemia (Blood and lymphatic system disorders) | 14 (20) | 1 (1) | 15 (19)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (5) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (6) | 1 (1) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 2 (2) | 11 (11)
Chorioretinopathy (Eye disorders) | 5 (7) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
MEK inhibitor-assessed serous retinopathy (Eye disorders) | 14 (15) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 1 (1) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 27 (37) | 4 (8) | 9 (11)
Diarrhoea (Gastrointestinal disorders) | 65 (111) | 10 (26) | 9 (10)
Dry mouth (Gastrointestinal disorders) | 12 (13) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 11 (11) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 48 (67) | 4 (5) | 7 (13)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 35 (44) | 3 (4) | 7 (8)
Asthenia (General disorders) | 12 (15) | 1 (1) | 11 (14)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 12 (13) | 2 (2) | 0 (0)
Fatigue (General disorders) | 42 (49) | 7 (7) | 5 (7)
Oedema (General disorders) | 2 (2) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 16 (20) | 3 (4) | 3 (3)
Peripheral swelling (General disorders) | 3 (3) | 1 (2) | 0 (0)
Pyrexia (General disorders) | 37 (47) | 1 (1) | 3 (8)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 6 (6) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 1 (1) | 4 (6)
Urinary tract infection (Infections and infestations) | 13 (14) | 1 (1) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (13) | 0 (0) | 4 (4)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (10) | 4 (6) | 5 (6)
Aspartate aminotrasferase increased (Investigations) | 10 (15) | 4 (4) | 6 (6)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 2 (3) | 4 (5)
Blood creatine phosphokinase increased (Investigations) | 25 (41) | 2 (3) | 5 (7)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 4 (5) | 1 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 7 (11) | 1 (4) | 9 (10)
Urine output decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 22 (23) | 2 (2) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 3 (3) | 2 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 7 (8) | 0 (0) | 7 (10)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (4)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (11) | 0 (0) | 5 (7)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (7) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (17) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (10) | 1 (1) | 9 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0) | 7 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 4 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 13 (14) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 6 (6) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (12) | 2 (2) | 14 (19)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 0 (0) | 4 (4)
Dysuria (Renal and urinary disorders) | 4 (4) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 0 (0) | 3 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 49 (62) | 7 (11) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 16 (19) | 4 (6) | 5 (7)
Rash (Skin and subcutaneous tissue disorders) | 31 (44) | 5 (5) | 6 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (18) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 0 (0) | 10 (13)
Hypotension (Vascular disorders) | 7 (9) | 1 (1) | 3 (7)
Chest pain (General disorders) | 0 (0) | 0 (0) | 3 (3)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (5)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 6 (8)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 5 (5)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 4 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (2) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 10 (12)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4)
Vitiligo (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 7 (11)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 6 (7)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 3 (7)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 4 (4)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pruritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 5 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or present ation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03178851/Prot_SAP_000.pdf